CLINICAL TRIAL: NCT01174212
Title: Effect of Prophylactic Antibiotics on Intra-Operative Culture Results
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Craig J Delle Valle, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10020102
Record Dates: First submitted 2010-07-27; First posted 2010-08-03 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Infection; Arthroplasty
Keywords: revision; infection; knee; hip; replacement; antibiotics
MeSH Terms: conditions — Infections | interventions — Second-Look Surgery; Arthroplasty; Anti-Bacterial Agents; Cefazolin; Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Patients receiving antibiotics approximately 1 hour prior to incision are considered to be in the experimental group of this study.
  Interventions: Procedure: Prophylactic Antibiotics
- Control (Other): Control group is to receive no antibiotics until the intraoperative cultures have been obtained.
  Interventions: Procedure: Control Antibiotics

INTERVENTIONS:
Procedure: Prophylactic Antibiotics — Preoperative Antibiotics
  Other Names: Revision; Arthroplasty; Infection; Antibiotics; Ancef; Vancomycin
  Arms: Experimental
Procedure: Control Antibiotics — Antibiotics will be held until intraoperative cultures have been obtained.
  Other Names: Arthroplasty; Infection; Antibiotics
  Arms: Control

SUMMARY:
Subjects will be consented and then determined randomly whether they will receive antibiotics prior to their surgery or during their surgery. Each patient will have cultures taken before and during their surgery from the infected hip or knee. Results will be compared after completion of the study.

DETAILED DESCRIPTION:
It is unknown whether giving pre-operative antibiotics affects the results of intraoperative bacterial cultures. This is an important question as antibiotics are often not given prior to surgery out of concern that accurate culture results will not be obtained. It is important to obtain accurate cultures so that targeted antibiotic therapy can be used. However, delaying the administration of antibiotics also delays the onset of treatment. Currently, the optimal course of action is unknown. The purpose of this study is to resolve this issue and determine if prophylactic antibiotics affect intra-operative culture results in patients undergoing revision hip or knee arthroplasty surgery for infection.

This is a prospective randomized clinical study to determine if prophylactic antibiotics affect intra-operative culture results in patients undergoing revision hip or knee arthroplasty surgery for infection. Pre-operatively, patients will have their affected joint aspirated and this fluid will be sent for cultures. Patients are then randomized to receive prophylactic antibiotics (Vancomycin and Ancef) within one hour prior to surgery or to have pre-operative antibiotics withheld. Every patient then has their affected joint cultured intra-operatively. All samples will be evaluated for the presence of aerobic bacteria, anaerobic bacteria, mycobacteria, and fungus. Pre-operative and post-operative cultures in both study populations are compared to determine the effects of pre-operative antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* prior arthroplasty surgery of the hip or knee
* presentation to clinic with infected joint
* scheduled for revision surgery

Exclusion Criteria:

* patients who have received antibiotics for any reason within 4 weeks of their pre-operative culture
* infected native joints
* septic patients
* refusal of participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in cultures obtained preoperatively and intraoperatively | 1 year
  Patients suspected of having an infected total hip or knee replacement in the post-operative period will be evaluated clinically. Preoperative and intraoperative revision cultures will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Rothman Institute, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Burnett RS, Aggarwal A, Givens SA, McClure JT, Morgan PM, Barrack RL. Prophylactic antibiotics do not affect cultures in the treatment of an infected TKA: a prospective trial. Clin Orthop Relat Res. 2010 Jan;468(1):127-34. doi: 10.1007/s11999-009-1014-4. Epub 2009 Aug 11. PMID 19669849